CLINICAL TRIAL: NCT06308666
Title: Performance of DAILIES TOTAL1 Daily Disposable Contact Lenses in Habitual Soft Lens Wearers Who Report Substantial Digital Device Use
Acronym: FOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46091
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Refit (Experimental): Refit and dispense participant with delefilcon A contact lenses and evaluate lens performance
  Interventions: Device: Delefilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Daily disposable silicone hydrogel contact lenses indicated for the optical correction of myopia and hyperopia
  Other Names: DAILIES TOTAL1®

SUMMARY:
The purpose of this study is to evaluate the performance of DAILIES TOTAL1 daily disposable contact lenses with regards to subjective symptoms (comfort, dryness, vision) in lens wearers who use identify themselves as substantial digital device users (at least eight hours of digital device use per day).

ELIGIBILITY:
Inclusion Criteria:

1. Are between 18 and 40 years of age (inclusive) and has full legal capacity to volunteer;
2. Have read and signed an information consent letter;
3. Are willing and able to follow instructions and maintain the appointment schedule;
4. Are a digital device user (at least 8 hours on a typical day using any combination of digital devices such as personal computer [PC], laptop, smartphone or tablet);
5. Are a habitual wearer of daily wear, spherical, soft contact lenses (no bifocal or multifocal contact lenses, no extended wear or monovision) for at least 5 days/week and at least 13+ hours/day on a typical day during the month prior to enrolment;
6. The habitual lens type brand will be restricted such that a maximum of 7 participants will be included in the study for each lens brand/material;
7. Have a vertex corrected spherical equivalent distance refraction within -0.50 Diopter (D) to -9.00D in each eye;
8. Have a vertex corrected refractive cylinder ≤ -0.75 cylindrical correction in each eye after vertexing to the corneal plane;
9. Demonstrate an acceptable fit and achieves best corrected visual acuity of at least 0.10 logMAR in each eye with DAILIES TOTAL1® contact lenses;
10. Are willing to wear DAILIES TOTAL1® contact lenses at least 5 days per week and 13+ hours per day throughout the study.

Exclusion Criteria:

1. Are participating in any concurrent clinical or research study involving intervention or invasive ocular tests;
2. Are presbyopic or habitually use a reading addition for close work;
3. Have any known active* ocular disease and/or infection; [* For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and mild dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.]
4. Meet the diagnosis of dry eye disease as per the following combination:

   1. Meets the symptom criteria of Contact Lens Dry Eye Questionnaire (CLDEQ-8) score ≥12
   2. And they show 1 of the following 2 signs:

      * Either sodium fluorescein (NaFl) staining (either [cornea >5 dots] or [conjunctiva >9 dots] or [lid margin >2mm length AND ≥25% width]);
      * Or non-invasive tear film break-up time (NITBUT) (no contact lens) <10 seconds.
5. Have a systemic condition that in the opinion of the investigator may affect a study outcome variable;+ [+ Any potential exclusion will be reviewed with the Lead Investigator or Principal Investigator prior to final decision making.]
6. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
7. Are a current wearer of DAILIES TOTAL1® daily disposable contact lenses;
8. Have known sensitivity to the diagnostic pharmaceutical sodium fluorescein to be used in the study;
9. Have undergone refractive error surgery;
10. Are a member of the Centre for Ocular Research & Education (CORE) directly involved in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between March 2024 and October 2024. The first participant was enrolled on March 18, 2024 and the last participant was enrolled on October 9, 2024.
Pre-assignment Details: Out of the 41 participants that were enrolled, 35 met the inclusion critieria, and 35 were dispensed with the study treatment.
Period: Overall Study
Arm/Group | Refit
Started | 35
Completed | 32
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Refit
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 35

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Comfort After 8 Hours or More of Digital Device Use
Description: Participants rate their overall comfort after 8 hours or more of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 14+2
Population: 3 people discontinued before the study could be completed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 96 [70 to 100]

2. Primary Outcome: Subjective Rating of Dryness After 8 Hours or More of Digital Device Use
Description: Participants rate their overall dryness after 8 hours or more of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 14+2
Population: 3 people discontinued before the study could be completed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 93 [50 to 100]

3. Primary Outcome: Subjective Rating of Clarity of Vision After 8 Hours or More of Digital Device Use
Description: Participants rate their overall clarity of vision after 8 hours or more of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 14+2
Population: 3 people discontinued before the study could be completed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [75 to 100]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Regular investigator assessment
Arm/Group | Refit
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT06308666/Prot_SAP_000.pdf